CLINICAL TRIAL: NCT03343041
Title: Pilot Study of Low-Carbohydrate Enteral Nutrition in Patients With Bacterial Septic Shock
Brief Title: Study of Low Carbohydrate Enteral Nutrition in Patients With Bacterial Septic Shock
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid and lack of resources
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000021424
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Bacterial Sepsis

STUDY DESIGN:
Intervention Model Description: The ultimate goal is to perform a prospective, single-center, double-blinded, parallel group, randomized, controlled trial on the safety and efficacy of low-carbohydrate enteral nutrition in adult patients admitted to the MICU with bacterial septic shock.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low carbohydrate nutrition (Active Comparator): We will use a low-carbohydrate nutrition (LCN) formulated by the MICU registered dietitian and pharmacy staff, who routinely prepare enteral and parenteral nutrition which will provide:
  5% carb, 41% protein, 54% lipid.
  Interventions: Dietary Supplement: low-carbohydrate nutrition
- standard enteral nutrition (Active Comparator): The standard enteral nutrition (SEN) and per cent contribution of carbohydrates used in the Yale MICU is as follows:
  Jevity 1.2 56% carb, 29.5% lipid, 18.5% protein Diabetisource 33% carb, 44% lipid, 20% protein Promote 55% carb, 25% lipid, 25% protein Vital AF 37% carb, 40% lipid, 25% protein Peptamin Intense 29% carb, 34% lipid, 37% protein Osmolite 1.5 54% carb, 29.5% lipid, 16.5% protein
  Interventions: Dietary Supplement: Standard enteral nutrition

INTERVENTIONS:
Dietary Supplement: low-carbohydrate nutrition — low-carbohydrate enteral nutrition
  Arms: low carbohydrate nutrition
Dietary Supplement: Standard enteral nutrition — standard enteral nutrition
  Arms: standard enteral nutrition

SUMMARY:
This pilot study aims to test the tolerability of low-carbohydrate enteral nutrition in patients with bacterial septic shock.

DETAILED DESCRIPTION:
This study seeks to assess the tolerability of utilizing low-carbohydrate nutrition in patients admitted to the MICU with bacterial septic shock. Low carbohydrate feeds have been used before in the critical care setting and were well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 admitted to the MICU with a diagnosis of severe sepsis or septic shock
2. Patients with 35 > BMI > 18.5
3. Patients with serum pro-calcitonin > 1 ng/mL in the first 24 hours of hospitalization

Exclusion Criteria:

1. Patients with chronic kidney disease as defined by glomerular filtration rate < 60 for > 6 months
2. Patients with chronic liver disease as defined by radiographic or tissue evidence of cirrhosis or persistently abnormal liver function tests for > 6 months
3. Patients with current malignancies
4. Patients with autoimmune disease on current immunotherapy
5. Patients on corticosteroids at doses of prednisone or prednisone-equivalents > 5 mg for > 6 months
6. Patients with weight-reduction surgeries
7. Patients with positive viral studies in the first 24 hours of admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Length of stay (LOS) in the ICU. | discharge: average 5 days.
  The primary clinical outcome will be to reduce the length of stay (LOS) in the ICU. Average length of stay is 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wang, MD PhD, Principal Investigator — Yale School of Medicine Department of Rheumatology
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States